CLINICAL TRIAL: NCT00176644
Title: Phase II Trial of Transdermal Estradiol in Patients With Hormone Refractory Prostate Cancer
Brief Title: Phase II Trial of Transdermal Estradiol for Hormone Refractory Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment ineffective
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445280; CINJ 080419 (Other: Cancer Institute of New Jersey); P30CA072720 (NIH); NCT00255632 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transdermal estradiol (Experimental)
  Interventions: Drug: Transdermal Estradiol

INTERVENTIONS:
Drug: Transdermal Estradiol — application of 4 transdermal estradiol patches, each patch releases a dose of 0.1 mg/day for a total dose of 0.4 mg/day. All four patches will be changed every 7 days. This continuous weekly schedule will be followed until the patient goes off-study.
  The patch will be applied to a clean, dry, intact area of the lower abdomen or the upper quadrant of the buttock. The sites should be rotated weekly. If a patch falls off during the 7 days, a new patch will be applied for the remainder of the 7 day period. At the end of the 7 days all four patches will be changed.

SUMMARY:
Multiple trials have shown the efficacy of estrogen therapy in metastatic prostate cancer, and most recently trials have supported the use of transdermal estrogens (patch) in the patient population with a decreased risk of cardiovascular disease as compared to the oral estrogens. We plan to study the use of transdermal estrogen at a dose of 0.4mg qd. We will evaluate the toxicities and measure quality of life. We will assess PSA response and measurable disease response. This will be a trial available to the Cancer Institute of New Jersey Oncology Group. We will enroll a total of 33 patients. We will plan to enroll 10 at CINJ.Patients will wear the patches (4) continuously. We will obtain blood work and clinic evaluations every three weeks. We will assess quality of life through a questionnaire given to patient every three weeks.

ELIGIBILITY:
Inclusion Criteria

* Patients with metastatic prostate adenocarcinoma, who have failed initial hormone therapy and who have had progression after at least one chemotherapy regimen that included docetaxel. Patients on antiandrogens must have progression after withdrawal of the antiandrogen for 4 weeks (flutamide) or 6 weeks (bicalutamide).
* PSA ≥ 10 ng/ml.
* Patients who have received LHRH agonist therapy for > 1 month must maintain agonist therapy while on-study. Patients who have not received agonist therapy or received < 1 month of therapy, may not begin or continue agonist therapy while on-study.
* Age >18 years and an estimated life expectancy of at least 4 months.
* ECOG performance status ≤ 2 (see Appendix B).
* Full recovery from the effects of any prior surgery or radiation therapy within 4 weeks of study entry.
* Serum creatinine ≤ 1.5 x ULN
* Total bilirubin < ULN
* Transaminases (SGOT and/or SGPT) ≤ 2 X institutional upper limit.
* Capacity to give informed, written consent.

Exclusion Criteria

* Any coexisting medical condition precluding full compliance with the study.
* Any history of deep venous thrombosis (DVT) or pulmonary embolus. Patients with a DVT on anticoagulants for ≥ 6 months will be eligible.
* Known CNS metastasis.
* The discontinuation of flutamide or bicalutamide < 4 or 6 weeks respectively.
* History of severe cardiovascular disease (AHA class III or IV; see Appendix C), uncontrolled CHF or life threatening cardiac dysrhythmia in the past 6 months.
* Herbal supplements may not be used while on-study and patients must have discontinued use for ≥ 1 week before entering on-study.
* Patients with a known hypersensitivity to estrogen.
* Triglyceride > 200 mg/dl.
* Prior estramustine.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (6):
- United States (6):
  - CentraState Healthcare System, Freehold, New Jersey
  - Robert Wood Johnson University Hospital/CINJ at Hamilton, Hamilton, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Overlook Hospital, Summit, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Cancer Institute of New Jersey (a comprehensive cancer center) and 4 community hospitals within the Cancer Institute of New Jersey Oncology Group from May 2005 through April 2008.
Groups:
- Transdermal Estradiol: Transdermal Estradiol : application of 4 transdermal estradiol patches, each patch releases a dose of 0.1 mg/day for a total dose of 0.4 mg/day. All four patches will be changed every 7 days. This continuous weekly schedule will be followed until the patient goes off-study.
  The patch will be applied to a clean, dry, intact area of the lower abdomen or the upper quadrant of the buttock. The sites should be rotated weekly. If a patch falls off during the 7 days, a new patch will be applied for the remainder of the 7 day period. At the end of the 7 days all four patches will be changed.
Period: Overall Study
Arm/Group | Transdermal Estradiol
Started | 23
Completed | 22
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With PSA Response
Description: PSA Response is a critical outcome measure used to assess the efficacy of treatments for conditions such as prostate cancer. PSA, or Prostate-Specific Antigen. The PSA Response is a measure of the change in PSA levels before and after a specific treatment intervention.
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 23
percentage of participants | 8.7

2. Secondary Outcome: To Measure Quality of Life of Participants Receiving Therapy With the Functional Assessment of Cancer Therapy-Prostate Scale (FACT-P).
Time Frame: 3 years
Population: Outcome Measure was pre-specified to be assessed based on achieving a certain pre-requisite response rate
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

3. Secondary Outcome: Measurable Disease Response Assessment in Participants With Hormone and Chemotherapy Refractory Prostate Cancer
Time Frame: 4 years
Population: Outcome Measure was pre-specified to be assessed based on achieving a certain pre-requisite response rate
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression
Time Frame: 3 years
Population: Outcome Measure was pre-specified to be assessed based on achieving a certain pre-requisite response rate
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

5. Secondary Outcome: Plateau Level of Estradiol and Testosterone Response in Androgen-Resistant Population With 0.4mg/Day Transdermal Estradiol Patch
Time Frame: 3 years
Population: Outcome Measure was pre-specified to be assessed based on achieving a certain pre-requisite response rate
Arm/Group | Transdermal Estradiol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years and 6 months
Arm/Group | Transdermal Estradiol
Serious Adverse Events (participants affected / at risk) | 5/23
Other Adverse Events (participants affected / at risk) | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Estradiol (N=23)
Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Pain - Bone (General disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstruction, GU - Urethra (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transdermal Estradiol (N=23)
Pain - Bone (General disorders) | 3 (3)
Pain - Breast (General disorders) | 3 (3)
Pain - Extremity-limb (General disorders) | 3 (3)
Pain - Back (General disorders) | 3 (3)
Pain - Neck (General disorders) | 2 (2)
Pain - Other (Specify, __) (General disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5)
Sweating (diaphoresis) (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 2 (2)
Calcium, serum-low (hypocalcemia) (Investigations) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 2 (5)
Edema: limb (Blood and lymphatic system disorders) | 3 (5)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Gynecomastia (Reproductive system and breast disorders) | 2 (2)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes